CLINICAL TRIAL: NCT05830591
Title: The Role of Gut-oral Axis Microbiome in Autism Spectrum Disorders
Brief Title: Gut-oral Axis Microbiome in Autism Spectrum Disorders
Status: Recruiting | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 20/21
Record Dates: First submitted 2023-03-29; First posted 2023-04-26 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Autism Spectrum Disorder; Microbiota
Keywords: Autism Spectrum Disorder; Microbiota; Inflammatory cytokines
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Oral swabs and fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Children with autism disorders 1-5 years: Children coming to the Division of Child Neurology and Psychiatry for the first clinical evaluation (1 year to 5 years old)
  Interventions: Other: Characterization of the microbiome in oral and fecal samples
- Children with autism disorders 6-17 years: Children with confirmed ASD diagnosis (6 years to 17 years old) coming to the Odonto-Stomatology Department for the periodical dental hygiene session
  Interventions: Other: Characterization of the microbiome in oral and fecal samples
- Children control group: Children with matched demographic characteristics accessing our Institute for different purposes
  Interventions: Other: Characterization of the microbiome in oral and fecal samples

INTERVENTIONS:
Other: Characterization of the microbiome in oral and fecal samples — The oral and fecal samples are collected during the periodical dental hygiene session at the odonto-stomatology unit and during day hospital for younger children admitted for the first clinical evaluation at Division of Child Neurology and Psychiatry. Procedures will follow standardized protocols.

SUMMARY:
Autism Spectrum Disorder (ASD) is a neurodevelopment disorder characterized by impairment in social interaction, communication, and behavior, as well as sensory challenges. In addition, secondary symptoms can appear, such as gastrointestinal disorders. Gut microbiota has an important role in the harvest of nutrients and energy from our diet. It influences a wide range of metabolic, developmental, and physiological processes such as the maintenance of the gut epithelial layer, immune system development, protection against pathogens, detoxification and xenobiotics degradation. The ecosystem of a healthy human gastrointestinal (GI) tract is mainly populated by Firmicutes and Bacteroidetes phyla, to a lesser extent by Actinobacteria and Proteobacteria, in this case the microbiota is in an eubiosis condition. Whether a disturbance of the microbial ecosystem occurs, gut microbiota is in a dysbiosis condition and it could lead different metabolic disorders. The two-way communication between gut microbiota and central nervous system (CNS) affects stress response, pain perception, neurochemistry and several disorders. The gut microbiota in ASD patients revealed some peculiarities such as the high percentage of Propionibacter and Clostridium, well known for their production of pro inflammatory metabolites, or an increment of Sutterella spp. and Ruminococcus torques, which are negatively associated with the health of the gut. Recent studies suggest that also the oral microbiota may be involved in ASD symptoms assuming the existence of a "microbiota-oral-brain axis". ASD patients are often suffering of several oral cavity disorders like caries, gingivitis and periodontitis, probably due to the poor oral hygiene. These disorders are linked to a dysbiosis of the oral microbiota: the characterization of the ASD subjects oral microbiota showed a lower biodiversity of bacteria species and different levels of specific bacteria, comparing to the controls. Several studies suggest that some bacteria species invade the blood-brain barriers as well as their metabolites, triggering inflammatory response and an alteration of the metabolic activity in the CNS. It has been demonstrated that ASD patients have a high level of pro-inflammatory cytokines and chemokines in the cerebrospinal fluid and an upregulation of the microglia. The oral microbiota could also affect the lower GI tract and have a significant role within the ASD-associated GI disorders and CNS inflammation

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a neurodevelopment disorder characterized by impairment in social interaction, communication, and behavior, as well as sensory challenges. In addition to the main symptoms, secondary symptoms can appear, such as gastrointestinal disorders. Gut microbiota has an important role in the harvest of nutrients and energy from our diet. Furthermore, it influences a wide range of metabolic, developmental, and physiological processes such as the maintenance of the gut epithelial layer, immune system development, protection against pathogens, detoxification and xenobiotics degradation. The ecosystem of a healthy human gastrointestinal (GI) tract is mainly populated by Firmicutes and Bacteroidetes phyla, to a lesser extent by Actinobacteria and Proteobacteria, in this case the microbiota is in an eubiosis condition. Whether a disturbance of the microbial ecosystem occurs, gut microbiota is in a dysbiosis condition and it could lead different metabolic disorders. For instance, the two-way communication between gut microbiota and central nervous system (CNS) affects stress response, pain perception, neurochemistry and several disorders. The gut microbiota in ASD patients revealed some peculiarities such as the high percentage of Propionibacter and Clostridium, well known for their production of pro inflammatory metabolites (like some short-chain fatty acids: acetate and propionate) or an increment of Sutterella spp. and Ruminococcus torques in feces of ASD children, which are negatively associated with the health of the gut. Similarly, very recent studies suggest that also the oral microbiota may be involved in ASD symptoms assuming the existence of a "microbiota-oral-brain axis". ASD patients are often suffering of several oral cavity disorders like caries, gingivitis and periodontitis, probably due to the poor oral hygiene. These disorders are linked to a dysbiosis of the oral microbiota: as a matter of fact, the characterization of the ASD subjects oral microbiota showed a lower biodiversity of bacteria species and different levels of specific bacteria, comparing to the controls. Several studies suggest that some bacteria species invade the blood-brain barriers as well as their metabolites, triggering inflammatory response and an alteration of the metabolic activity in the CNS. Interestingly, it has been demonstrated that ASD patients have a high level of pro-inflammatory cytokines and chemokines in the cerebrospinal fluid and an upregulation of the microglia. The oral microbiota could also affect the lower gastro-intestinal (GI) tract, given the transit of bacteria from the oral cavity to the gut, leading to different effects depending on the type of bacteria. This implies that an oral microbiota dysbiosis may be one of the leading causes of the gut microbiota dysbiosis reported in numerous ASD studies as demonstrated by studies of the Human Microbiome Project, the 45% of the gut and oral microbiota bacteria over-lap. In light of these facts, the oral microbiota could have a significant role within the ASD-associated GI disorders and CNS inflammation. The main objective of this project is to identify descriptive features relative to bacterial species in gut and oral microbiota of pediatric subjects with ASD diagnosis. The purpose is to find whether these species overlap in order to identify descriptive features of ASD, which are collectable by means of a simple oral swab (rather than a fecal sample). These species will be identified with both DNA sequencing, followed by bioinformatic analysis, and a culturomic approach. The innovative approach of "network analysis" will be employed in order to find definite bacterial consortia, named Species Interacting Groups (SIGs) able to collect the abovementioned featuring species. These data could be useful for a better ASD description in terms of bacterial compositional differences, especially within a defined pediatric group.

ELIGIBILITY:
INCLUSION CRITERIA

Case group

1. Caucasian
2. Diagnosed with ASD or with a newly formulated diagnosis of ASD
3. Aged between 1 and 17 years

Control group

1. Caucasian
2. Healthy at the time of sampling
3. No ASD or other neurological disorders
4. Aged between 1 and 17 years

EXCLUSION CRITERIA

1. Antibiotic use in the month before sample collection
2. Probiotic use in the month before sample collection
3. Other neurological diseases
4. Chronic inflammatory diseases
5. The use of constipation drugs during the three days before sample collection

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric subjects:
  * children coming to the Division of Child Neurology and Psychiatry for the first clinical evaluation (1 year to 5 years old)
  * children with confirmed ASD diagnosis (6 years to 17 years old) coming to the Odonto-Stomatology Department for the periodical dental hygiene session.
  * children control group with matched demographic characteristics accessing our Institute for different purposes
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To compare oral and GI microbiota | At baseline
  Oral and GI bacterial species will be evaluated in oral and fecal samples collected and compared through bioinformatic and statistical analysis among case and control groups to isolate the discriminant ones. The technical activity is focused on samples DNA extraction and sequencing and on a culturomic approach.

SECONDARY OUTCOMES:
To evaluate the association between the key bacteria species found in ASD microbiota and soluble concentration of salivary cytokines | At baseline
  Oral and GI bacterial species will be evaluated in oral and fecal samples. The soluble concentrations (picograms per millilitre) of a panel of 27 cytokines and chemokines will be simultaneously assessed in saliva samples.
To evaluate the association between the key bacteria species found in ASD microbiota and soluble concentration of salivary chemokines | At baseline
  Oral and GI bacterial species will be evaluated in oral and fecal samples. The soluble concentrations (picograms per millilitre) of a panel of 27 cytokines and chemokines will be simultaneously assessed in saliva samples.
To evaluate the association between the microbiota structure and the severity of the ASD symptoms | At baseline
  Oral and GI bacterial species will be evaluated in oral and fecal samples. Clinical data will be collected from medical records.
To evaluate the association between the microbiota structure and eating habits of ASD children | At baseline
  A food diary will be distributed at enrollment to evaluate eating habits of ASD children

CONTACTS AND LOCATIONS:
Overall Officials: Manola Comar, BSc, Study Director — Institute for Maternal and Child Health IRCCS Burlo Garofolo
Locations (1):
- Institute for Maternal and Child Health - IRCCS "Burlo Garofolo", Trieste, Italy

IPD SHARING:
Plan to Share IPD: Undecided